CLINICAL TRIAL: NCT06608082
Title: Study of the Vascularization of the Vaginal Slice After Total Laparoscopic Hysterectomy, Using Indocyanine Green Injection. Prospective Feasibility Study
Brief Title: Study of the Vascularization of the Vaginal Slice After Total Laparoscopic Hysterectomy, Using Indocyanine Green Injection.
Acronym: HYSTINDO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOI 2023 CHAUVET
Record Dates: First submitted 2024-08-23; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Hysterectomy; Vascularization; Complication of Surgical Procedure
Keywords: indocyanine green; laparoscopic hysterectomy; Post-operative complications of hysterectomy; TRACKER software; imaging technique
MeSH Terms: conditions — Neovascularization, Pathologic

STUDY DESIGN:
Intervention Model Description: Study the presence of indocyanine green in the vaginal cuff during the total laparoscopic hysterectomy, in order to assess intraoperative vascularization of the area (fluorescence intensity value different from 0). This is a prospective feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Totale hysterectomy with indocyanine green and fluorescence intensity analysis (Other): Patient scheduled to undergo total hysterectomy through a surgically accessible laparoscopic procedure.
  The difference from standard care is that during the intraoperative period, at the end of the procedure, the patient will receive a diluted bolus of indocyanine green. The collected images will be analyzed using the TRACKER software in order to assess intraoperative vascularization of the area (fluorescence intensity value different from 0).
  Interventions: Diagnostic Test: indocyanine green injected intravenously

INTERVENTIONS:
Diagnostic Test: indocyanine green injected intravenously — During the procedure, after performing the hysterectomy, indocyanine green will be injected intravenously into the patient. A fluorescence video of the vaginal cuff will be recorded. The fluorescence of the recorded images will be analyzed by fluorescence analysis software to obtain an objective value of fluorescence.

SUMMARY:
Hysterectomy is one of the most common surgical procedures in gynecology, especially by laparoscopy. Post-operative complications of hysterectomy are numerous and their causes are poorly understood.

Indocyanine green is a fluorescent dye that, when exposed to infrared light, makes it possible to visualize the vascularization by fluorescence.

The project consists in studying the vascularization of the vaginal cuff after total laparoscopic hysterectomy using the injection of indocyanine green. This is a prospective feasibility study.

During the procedure, after performing the hysterectomy, indocyanine green will be injected intravenously into the patient. A fluorescence video of the vaginal cuff will be recorded. The fluorescence of the recorded images will be analyzed by fluorescence analysis software to obtain an objective value of fluorescence. The fluorescence values will be compared to the occurrence or absence of postoperative complications.

This is the first study using this imaging technique combined with indocyanine green in this surgery. This study will employ a novel objective sequential fluorescence analysis software that has already proven its effectiveness in digestive surgery. The sequential measurement of the change in fluorescence intensity visualized in the images of laparoscopy will enable the production of vaginal perfusion graphs using a video modeling tool such as the TRACKER software. This software measures the evolution of green levels in a region of interest, from which a time-fluorescence curve can be obtained. The presence of fluorescence will be defined by a fluorescence intensity value of Fmax-Fmin on the graph.

DETAILED DESCRIPTION:
To perform this study, the patient will undergo a preoperative consultation with a senior surgeon and an anesthetist from the department to schedule the surgical procedure and discuss potential inclusion in the protocol.

Day before the surgery : The patient will give an informed and written consent and will be enrolled in the study.

The day of the intervention : The planned surgical procedure will be performed as initially scheduled by the surgeon (total hysterectomy). The difference from standard care is that during the intraoperative period, at the end of the procedure, the patient will receive a diluted bolus of indocyanine green (25 mg in 10 ml of 5% glucose solution), at a dose of 0.2 mg/kg. Subsequently, the laparoscopic camera system will be switched to an infrared camera system to visualize intra-abdominal fluorescence using the trocars used during the surgery. A video recording sequence of the vaginal cuff, lasting two to five minutes, starting from the moment of the indocyanine green injection will be collected by the investigator. The collected images will be analyzed using the TRACKER software (Douglas Brown, Open Source Physics, Boston MA, USA).

Postoperative period : A postoperative consultation will take place between 3 and 8 weeks after the surgery with one of the senior physicians from the department. Postoperative progress and early complications (dehiscence, cuff infection, abscess, or hematoma) will be documented, along with anatomopathological examination data and the final diagnosis.

The postoperative follow-up will remain consistent with the usual protocol following this procedure. The protocol does not involve any additional visits, thus no potential extra coast.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient scheduled to undergo total hysterectomy through a surgically accessible laparoscopic procedure.
* Patiente capable of providing informed consent to participate in the study.
* Patiente covered by the Social Security system.

Exclusion Criteria:

* Protected patient, under guardianship, curatorship or legal protection.
* Patient's refusal or inadequate understanding of the French language.
* Known allergy to iodine.
* Ongoing pregnancy and breastfeeding.
* Procedure requiring the use of indocyanine green.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-09-21 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Study the presence of indocyanine green in the vaginal cuff during the total laparoscopic hysterectomy, in order to assess intraoperative vascularization of the area (fluorescence intensity value different from 0). | 2 months
  An objective measurement of fluorescence will be employed. Sequential measurement of fluorescence intensity changes observed in the laparoscopy images will enable the creation of vaginal perfusion graphs using a video modeling tool like the TRACKER software (Douglas Brown, Open Source Physics, Boston MA, USA). This software tracks the evolution of green levels within a region of interest, from which a time-fluorescence curve can be derived.
  The presence of fluorescence will be defined by the fluorescence intensity value Fmax-Fmin. All procedures will be recorded and subsequently collected by the investigator. All collected images will undergo analysis using the TRACKER software (Douglas Brown, Open Source Physics, Boston MA, USA).

SECONDARY OUTCOMES:
Examine the different parameters derived from the perfusion curve. | 2 months
  The different parameters derived from the perfusion curve: minimum fluorescence intensity (Fmin), maximum fluorescence intensity (Fmax), difference in fluorescence intensity (Fmax-min), slope of fluorescence intensity, time ratio (TR).
Compare the objective fluorescence measurements to the surgeon's assessment. | through study completion, an average of 1 year
  Objective fluorescence measurements and surgeon's assessment (Likert scale). The uptake of fluorescence in the vaginal cuff and its intensity will be evaluated by the surgeon during the procedure using a Likert scale. The presence of fluorescence will be defined by a score from 0 to 4. The obtained score will be compared to the objective measurements of the fluorescence curve.
Evaluate the immediate or delayed tolerance of indocyanine green. | through study completion, an average of 1 year
  Side effects and occurrence of adverse events related to the injection of indocyanine green.
Assess the additional time added to the total operative duration by the protocol. | 2 months
  The time added to the total operative duration by the protocol. The duration of the phase corresponding to the protocol will be equal to the time between the injection of indocyanine green and the cessation of video recording in minutes. The total operative duration will be equal to the time between the incision time and the closure time in minutes.
Compare the vascularization of the vaginal cuff to patient characteristics. | 2 months
  Patient characteristics :IMC, age, tabacco consumption (yes/no), ASA score, gestation/parity, medical and surgical history, comorbidities, surgical indication, preoperative imaging (echography and/or MRI (yes/no) and conclusion), concomitant treatment, sexual activity (yes/no).
Compare the vascularization of the vaginal cuff to Surgical technique | 2 months
  Surgical technique : instrument and coagulation mode, energy type, suture type, thread type
Compare the vascularization of the vaginal cuff to Type of camera | 2 months
  Type of camera : SPIES, RUBINA, and FIREFLY systems
Compare the vascularization of the vaginal cuff to Post-operative complications | 2 months
  Post-operative complications : bleeding, fever, biological inflammatory syndrome, pain, early post-operative abscess, hemoperitoneum, hematoma, infection/abscess, fistula
Compare the vascularization of the vaginal cuff to State of the vaginal cuff | 2 months
  State of the vaginal cuff : Presence of visible sutures, On speculum examination : complete healing, ongoing healing, presence of dehiscence (size, time of occurrence) or evisceration and On vaginal palpation : presence or absence of dehiscence (size, time of occurence)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No